CLINICAL TRIAL: NCT00621738
Title: Effect of Mental Stress on Platelet Function in Healthy Subject
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Prof Georg Noll, University of Zurich
Other Study IDs: 1382
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: mental stress; cardiovascular risk factor; platelet adhesion
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Psychological stress is an independent cardiovascular risk factor. Activation of platelets plays an important role in atherosclerosis development and it could one of the mechanisms linking psychological stress and cardiovascular diseases

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects
* No smokers
* Written informed consent

Exclusion criteria:

* Smoking
* Alcohol- or Drug Abuse
* Pregnancy
* Use of benzodiazepins, Aspirin or NSAIDs in the last week before inclusion
* Participation to another study within the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, aging 18-80 years
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Georg Noll, MD, Principal Investigator — Cardiovascular Center Cardiology University Hospital Zurich
Locations (1):
- Cardiovascular Center Cardiology Univeristy Hospital of Zurich, Zurich, Switzerland